CLINICAL TRIAL: NCT01283191
Title: Using Behavioral Incentives to Promote Exercise Compliance in Cocaine Dependent Women
Brief Title: Behavioral Incentives to Increase Exercise in Cocaine Dependent Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD301598 1R36DA030619-01; R36DA030619 (NIH)
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Cocaine Dependence
Keywords: substance use; drug use; drug abuse; exercise; physical activity
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Incentives (Experimental): Vouchers for complying with target behavior
  Interventions: Behavioral: Behavioral Incentives
- Education Control (Placebo Comparator): Education class
  Interventions: Behavioral: Education Control

INTERVENTIONS:
Behavioral: Behavioral Incentives — Vouchers for complying with target behavior of treadmill walking
  Arms: Behavioral Incentives
Behavioral: Education Control — Education class
  Arms: Education Control

SUMMARY:
While physical activity has been associated with decreased craving and increased abstinence rates in smokers, few published studies have examined the effects of exercise on recovery from other drugs such as cocaine. One factor that has impeded such research has been low levels of patient compliance with exercise protocols. One robust strategy for promoting and maintaining behavior change is contingency management or Behavioral Incentives (BI). BI delivers incentives (prizes, vouchers) contingent upon target behaviors such as cocaine abstinence (Higgins et al., 1994); treatment attendance (Svikis et al., 1997) and other pro-social behaviors (Kirby et al., 1998). While the literature is replete with studies demonstrating the benefit of BI compared to control conditions (Stitzer & Petry, 2006), the translation of BI methods from research to clinical practice has met with some resistance. Contributing factors include philosophical differences (e.g., counselors feel extrinsic reinforcement undermines recovery) and practical barriers (e.g., monetary costs of incentives may be prohibitive). The latter concern was addressed by Petry (2005) who developed the "fish bowl" method, which uses escalating variable ratio procedures to reduce per patient costs of BI with similar effect sizes.

As a Stage 1 behavioral therapies development grant (Rounsaville et al., 2001), the primary aim of this research is to pilot test a BI intervention designed to promote regular physical activity in a sample of women receiving inpatient treatment for SUDs. The target behavior, physical activity, will be objectively defined as 30 minutes of observed treadmill walking at any intensity 3 days/week at Level 1, and 30 minutes of higher intensity physical activity that meets ACSM criteria for moderate exercise Level 2. Specifically, a pilot randomized clinical trial will compare rates of physical activity over a 6 week study period in a sample of N=50 women with Cocaine Dependence. All participants will complete baseline assessment, attend a 45-min Health and Fitness (HF) education group, followed by random assignment to either the experimental (BI) or control (C) groups, with equal daily access to on-site treadmills. Those randomized to BI, however, will also be eligible 3 days/week, to receive incentives for completing 30 minutes of treadmill walking.

Incentives will be dispensed using Petry Fish Bowl methods. Women assigned to the BI group will receive behavioral incentives (in the form of gift cards or prizes) for completing their scheduled exercise sessions (Level 1), and have the opportunity to earn "bonus" draws for meeting moderate intensity exercise criteria, as specified by ACSM (2007, revised) guidelines (Level 2). In Level 1, the number of tokens participants can draw from the gym bag (present study equivalent to "fishbowl") at each visit will be linked to exercise session attendance, with consistent attendance resulting in greater number of draws. In Level 2, the number of tokens a participant can draw from the gym bag will be linked to the intensity of the participant's exercise. Specifically, beginning in Week 2 of the study, participants will be re-evaluated for exercise capability. Those who pass the safety screen will be encouraged to exercise at a higher intensity, and those who do not will be re-evaluated until they obtain safety clearance. Once cleared, if the participant meets criteria for moderate exercise during her scheduled session, then she will be allotted a "bonus" draw (Level 2) for meeting Level 2 criteria, in addition to the escalating number of draws she would received for scheduled exercise session completion (Level 1).

Scheduled treadmill walking will be monitored and recorded for both BI and C group women. Follow-ups will occur at study midpoint and completion (3 and 6 weeks post-randomization, respectively), and at 4 weeks post-discharge. Assessments will focus on drug craving, mood, stress, motivation/self-efficacy, and physical health and well being. The investigators hypothesize that women in the BI group will complete more treadmill sessions and spend more time treadmill walking than those in the C group. As a Stage 1b therapy development RCT, study data will be used for effect size estimation in preparation for Stage 2 RCT. This dissertation proposal will provide benchmark data on the utility of BI for promoting physical activity. Further, it will promote exercise compliance, allowing scientists to better evaluate potential benefits of physical activity on treatment outcomes in women with SUDs.

ELIGIBILITY:
Inclusion Criteria:

* 1) at least 18 years of age
* 2) female
* 3) meet DSM-IV criteria for Cocaine Dependence (current)
* 4) medically cleared by the Rubicon staff physician to participate in a regular exercise program
* 5) able to provide informed consent for study participation.

Exclusion Criteria:

* 1)are pregnant
* 2)present with cognitive impairment, psychiatric instability, or language barriers that limit their ability to provide informed consent and participate in research assessments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Time in core sessions | 6 weeks
  Time (minutes) spent treadmill walking over 18 core sessions
Total time | 10 weeks
  Total time (minutes) spent treadmill walking over the 6 week study period (core sessions + additional sessions)

SECONDARY OUTCOMES:
Higher intensity time | 6 weeks
  Time (minutes) spent in higher intensity physical activity over 18 core sessions
Higher intensity total time | 6 weeks
  Total time (minutes) spent in higher intensity physical activity over the 6 week study period
Session number | 6 weeks
  Number of 30-minute treadmill sessions completed
Total session number | 6 weeks
  Number of total treadmill sessions (any duration)
Number of moderate sessions | 6 weeks
  Number of treadmill sessions at moderate intensity exercise
Total walking time | 6 weeks
  Total time walking on treadmill
Consecutive exercise sessions | 6 weeks
  Number of consecutive exercise sessions completed (3 days/week X 6 weeks)
Post-discharge exercise | 4 weeks
  Quantity and frequency of exercise during 4-week post-discharge follow-up
Relapse to drug use | 10 weeks
  Relapse to cocaine and other drug use post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Leila Z Islam, M.S., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Rubicon, Inc., Richmond, Virginia, United States